CLINICAL TRIAL: NCT06360003
Title: "Right Ventricular Outflow Tract Posterior Septum Pacing" in Predicting Ventricular Outflow Tract Ventricular Tachycardia Origin: a Single-center, Prospective, Single Blind, Randomised Controlled Study
Brief Title: "Right Ventricular Outflow Tract Posterior Septum Pacing" in Predicting Ventricular Outflow Tract Ventricular Tachycardia Origin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2024-01-109
Record Dates: First submitted 2024-03-28; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Ventricular Outflow Tract Ventricular Arrhythmias; Radio Frequency Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right Ventricular Outflow Tract (RVOT) Posterior Septum Pacing Group (Active Comparator)
  Interventions: Procedure: Right Ventricular Outflow Tract Posterior Septum Pacing
- Convention Group (Active Comparator)
  Interventions: Procedure: systemic mapping and ablation

INTERVENTIONS:
Procedure: Right Ventricular Outflow Tract Posterior Septum Pacing — The Right Ventricular Outflow Tract (RVOT) posterior septum pacing is routinely performed to observe the QRS complex characteristics of the 12 lead ECG (with a focus on comparing their differences with the R-wave amplitude of spontaneous ventricular arrhythmias in the right chest (V1~V3) leads). When the pacing-induced R-wave amplitudes are all lower than spontaneous VAs in V1~V3, we predict the origin of Left Ventricular Outflow Tract (LVOT), mapping and ablation in LVOT; otherwise we predict the origin of RVOT, mapping and ablation in RVOT.If fails, go to the opposite site to do mapping and ablation. If still fails, go to distal great cardiac vein (DGCV) to do mapping and ablation.
  Arms: Right Ventricular Outflow Tract (RVOT) Posterior Septum Pacing Group
Procedure: systemic mapping and ablation — The TC or ST ablation catheter is delivered to ventricular outflow tract (VOT) to perform systemic mapping and ablation.
  Arms: Convention Group

SUMMARY:
The goal of this clinical trial is to make clear that a new method, right ventricular outflow tract (RVOT) posterior septum pacing, has a greater accuracy in predicting the origin of ventricular outflow tract (VOT) ventricular arrhythmias (VAs) compared to the previous electrocardiographic standards for the identification of the origin of ventricular outflow tract. The secondary aim is to investigate, by using the new method, if it can optimize the procedure of radiofrequency catheter ablation.

Researches will break the method of this investigation into two steps:

First step have enrolled 100 patients. This step would be used to compare the results predicted by right ventricular outflow tract posterior septum pacing, with the previously used electrocardiographic criteria and actual target site.

The second step will enroll another 100 patients. In this step, patients will be divided into two groups, one being the new protocol group and the other being the convention group. Patients will also be followed up, for 1 month and 3 months at outpatient clinic post procedure. Procedure time, success rate, fluoroscopy exposure time and complications, are compared between RVOT posterior septum pacing group and convention group.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent form
* Age more than 18 years old
* Able to understand the purpose of the experiment, voluntarily participate, willing to complete follow-up according to the requirement of the experimental protocol.

Exclusion Criteria:

* Severe cardiopulmonary, liver and kidney dysfunction, and inability to tolerate surgery due to coagulation dysfunction
* Viral myocarditis, myocardial infarction or stroke with a course of less than six months
* Simultaneously accompanied by malignant tumours, with an expected lifespan of less than or equal to 1 year
* Severe thoracic deformity
* Advanced age (more than 90 years old)
* Other situations that the researcher deems unsuitable for participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Immediate Ablation Success | At the end of the first procedure
  Immediate Ablation Success is determined by the disappearance of ventricular arrhythmia after ablation, that cannot be induced by electrical stimulation and intravenous infusion of isoproterenol.
Rate of Ablation Complication | At the end of the first procedure
  Complications like cardiac tamponade, artery damage
Accuracy of RVOT posterior septal pacing protocol | At the end of the first procedure
  Target site predicted by RVOT posterior septal pacing protocol compared with actual target site and previous ecg criteria

SECONDARY OUTCOMES:
Incidence of Complications Post-operative | period of post-operative to hospital discharge, within 7 days
  Complications like cardiac tamponade, artery damage
Incidence of Complication | 1 months after first procedure
  Complications like pericardial effusion, pseudo arterial aneurysm
Rate of Recurrence during Follow up | 1 months after first procedure
  Recurrence of the ventricular arrhythmia during the follow up period after catheter ablation procedure
Incidence of Complication | 3 months after first procedure
  Complications like pericardial effusion, pseudo arterial aneurysm
Rate of Recurrence during Follow up | 3 months after first procedure
  Recurrence of the ventricular arrhythmia during the follow up period after catheter ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Zheng, PhD, Principal Investigator — Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University
Locations (1):
- Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China